CLINICAL TRIAL: NCT05337943
Title: Feasibility of Cognitive Behavioral Therapy vs. Bright Light Therapy to Treat Insomnia and Fatigue: an RCT
Brief Title: Cognitive Behavioral Therapy and Light Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 850360
Record Dates: First submitted 2022-04-13; First posted 2022-04-20 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Hypertension; Insomnia; Fatigue
MeSH Terms: conditions — Hypertension, Pulmonary; Sleep Initiation and Maintenance Disorders; Fatigue | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Behavioral Therapy-Insomnia (CBT-I) (Experimental): CBT-I treatment will receive 1 session every week, for 8 weeks (8 total sessions). The CBT-I sessions will be provided by a pool of clinical PhD psychology students by a trained professional. Each visit will be conducted via telehealth. Sessions will include discussions regarding such topics as sleep restriction, stimulus control and sleep hygiene. Review of sleep diaries will occur during the sessions.
  Interventions: Behavioral: CBT-I
- Bright Light Therapy (Experimental): Bright Light treatment will consist of 8 weeks of daily use of the Re-timer device. The Re-timer is worn like a pair of glasses and contains light emitting diodes mounted on the lower portion of the frame. The Re-timer emits blue-green 500 nm light with an intensity of ~500 lux lm/m2. Subjects will be instructed to use the device for 30 minutes within two hours of waking, in the morning on the full brightness setting.
  Interventions: Device: Bright Light Therapy
- Standard Care (No Intervention): Subjects will continue the care they routinely receive.

INTERVENTIONS:
Behavioral: CBT-I — Weekly sessions with a therapist to improve sleep for 8 weeks.
  Arms: Cognitive Behavioral Therapy-Insomnia (CBT-I)
Device: Bright Light Therapy — Daily light therapy for 30 minutes for 8 weeks.
  Arms: Bright Light Therapy

SUMMARY:
Cognitive behavioral therapy (CBT-I) is a common treatment for insomnia that does not use medications. While CBT-I is effective for insomnia, it does not tend to improve the waking symptom of fatigue. Another treatment, Bright Light Therapy, is used for treating seasonal depression and sleep disorders, and may improve fatigue and physical activity in individuals with PAH. The purpose of this study to assess the effects of Bright Light Therapy compared to CBT-I to treat insomnia and fatigue in patients with PAH.

DETAILED DESCRIPTION:
In a single site, 3-arm (Cognitive Behavioral Therapy [CBT-I] group; Bright Light Therapy group; Standard of Care group), parallel, randomized controlled trial we will enroll 36 subjects (n=12 per group) to assess the feasibility of Bright Light Therapy compared to CBT-I in subjects with pulmonary arterial hypertension (PAH) to treat insomnia (difficulty initiating sleep or maintaining sleep) and fatigue.

* To assess the recruitment and retention rates of CBT-I and Bright Light Therapy.
* To compare the effects of CBT-I and Bright Light Therapy to Standard of Care on (insomnia and fatigue severity) and secondary (wake after sleep onset and sleep onset latency) outcomes.
* To test the effects of CBT-I and Bright Light Therapy to Standard of Care on the secondary outcome physical activity.
* To test the effects of CBT-I and Bright Light Therapy to Standard of Care on the secondary outcomes: depression, dyspnea and QOL.

ELIGIBILITY:
Inclusion Criteria:

* PAH diagnosis
* Insomnia
* Fatigue

Exclusion Criteria:

* Untreated obstructive sleep apnea
* Subjects with left-sided valvular disease
* Hospitalized or acutely ill
* Any eye disease such as, but not limited to, cataracts, glaucoma, retinal disorders (e.g. macular degeneration), or previous eye surgery
* Subjects with photosensitivity (e.g. epilepsy)
* Manic-depressive psychosis or Bipolar Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lea Ann A Matura, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Behavioral Therapy-Insomnia (CBT-I) | Bright Light Therapy | Standard Care
Started | 1 | 3 | 2
Completed | 0 | 1 | 2
Not Completed | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy-Insomnia (CBT-I) | Bright Light Therapy | Standard Care | Total
Number analyzed (Participants) | 1 | 3 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (0) | 48.3 (17.8) | 55.0 (21.2) | 52.3 (15.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 1 | 2 | 1 | 4
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 3 | 2 | 6
Enrollment Arms [Count of Participants; unit: Participants] | 1 | 3 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Retention Rate
Description: Number of participants who completed all study procedures.
Time Frame: 8 weeks
Population: The participant randomized to CBT-I withdrew from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitive Behavioral Therapy-Insomnia (CBT-I) | Bright Light Therapy | Standard Care
Number analyzed (Participants) | 1 | 3 | 2
Participants | 0 | 1 | 2

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Cognitive Behavioral Therapy-Insomnia (CBT-I) | Bright Light Therapy | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT05337943/Prot_SAP_000.pdf